CLINICAL TRIAL: NCT07070102
Title: Population Pharmacokinetics of Temocillin in Acute Enterobacterial Pyelonephritis in Children
Acronym: TEMOKID-POP
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241684; 2025-A00368-41 (Registry Identifier: IDRCB ANSM)
Record Dates: First submitted 2025-06-23; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Pyelonephritis
Keywords: temocillin
MeSH Terms: conditions — Pyelonephritis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 blood samples of 1 mL. The study is observational because participants get these blood samples as part of routine medical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood samples — 2 blood samples of 1 mL

SUMMARY:
Temocillin, a 6-alpha-methoxypenicillin derivative of ticarcillin, is a narrow-spectrum antibiotic, primarily restricted to Enterobacterales. Therefore, its prescription for the treatment of febrile urinary tract infections requiring hospitalization in pediatrics appears interesting.

However, and despite marketing authorization in pediatrics for the treatment of complicated urinary tract infections (including acute pyelonephritis), the pharmacokinetic parameters of this antibiotic have not been specifically evaluated in pediatrics, and the optimal dose is not known in this population.

Through this study, we propose to determine the pharmacokinetic parameters of temocillin in children aged 0-15 years with a febrile urinary tract infection due to Gram-negative rod (GNR), without sepsis but requiring hospitalization. The results will help to establish dose recommendations for temocillin in the pediatric population, based on age and renal function.

DETAILED DESCRIPTION:
Clinical Context of Temocillin Use:

Temocillin is an old antibiotic, a 6-alpha-methoxypenicillin derivative of ticarcillin, which has been rediscovered in recent years due to its narrow spectrum of activity and its ability to resist hydrolysis by most beta-lactamases, including ESBL. Temocillin is bactericidal, is not impacted by the inoculum effect, and has a low selection of resistant mutants. Due to its narrow spectrum (essentially limited to Enterobacterales), it appears to have a reduced overall impact on the fecal microbiota.

Studies have retrospectively reported clinical and microbiological efficacy of temocillin in urinary tract infections caused by ESBL-producing Enterobacterales in children and adults.

More generally, Enterobacterales have a high susceptibility to temocillin, with susceptibility rates exceeding 90-95% in several epidemiological studies in both children and adults. This is higher than that of third-generation cephalosporins, which still remain the first-line treatment in recent french guidelines (GPIP, SPILF), As a result, temocillin has been approved for the treatment of acute pyelonephritis (febrile urinary tract infections), including in the pediatric population. In France, it is primarily used for the treatment of ESBL-associated febrile urinary tract infections.

Since september 2024, Robert Debré University Hospital uses temocillin has an empiricial antibiotic therapy for hospitalized cases of febrile urinary tract infections, without any sign of sepsis, at the recommended high dose of 50 mg/kg/day in 2 intravenous injections of 30 min spaced 12 hours apart.

Pharmacokinetic Data of Temocillin:

Temocillin is a bactericidal antibiotic for parenteral use, belonging to the beta-lactam family. Temocillin binds strongly to plasma proteins (approximately 80% binding) and has a prolonged elimination half-life of approximately 5 hours. Its elimination is primarily renal.

As with other beta-lactams, the best pharmacokinetic/pharmacodynamic (PK/PD) criterion correlated with the efficacy of temocillin appears to be the cumulative percentage of time over 24 hours during which temocillin's free concentration exceeds the minimum inhibitory concentration (fT>MIC) at steady state. A target fT>MIC 40% of is associated with antibacterial effect and in vivo survival.

In adults, Monte Carlo pharmacokinetic simulations have demonstrated that an IV regimen of 2 grams every 12 hours allows a %ft>MIC of 40% to be achieved in 95% of treated patients and for MICs up to 8 mg/L.

In children up to 15 years of age, the standard recommended dosage is 25 mg/kg/day in 2 IV injections (max. 4g/day) but a higher dosage of 50 mg/kg/day in 2 IV injections (max. 4g/day) is indicated for the treatment of severe infections (including acute pyelonephritis requiring hospitalization). However, these proposed regimens recommendations do not originate from paediatric PK/PD studies but are derived from adult studies. To date, no study has evaluated the pharmacokinetic parameters of temocillin specifically in children (<15 years), and the optimal dosage regimen maximizing the probability of reaching the target PK/PD criterion (fT>MIC of 40%) in the treatment of febrile urinary tract infections due to GNR is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 0 to 15 years
* Presenting with a febrile urinary tract infection due to GNR (a febrile urinary tract infection is defined as a urine culture showing significant leukocyturia (≥104) and direct examination showing GNR, in a patient with fever)
* Requiring hospitalization in the general pediatrics, emergency (short-stay hospitalization unit), nephrology, or intensive care units of the Robert-Debré University Hospital for a presumed period of at least 48 hours.
* Non-opposition of the legal representatives obtained by one of the investigator

Exclusion Criteria:

* Presence of sepsis (Phoenix score ≥ 2)
* Gram-positive cocci (GPC) urinary tract infection (Urinalysis before antibiotic therapy revealed significant leukocyturia (≥104) and direct examination revealed GPC)
* Known allergy to beta-lactam antibiotics
* Severe renal impairment (glomerular filtration rate <30 mL/min*1.73 m2)

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient aged 0 to 15 years (inclusive) presenting with a febrile urinary tract infection with BGN requiring hospitalization in the departments of the Robert-Debré University Hospital for a duration of at least 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Achievement of the theoretical PK/PD target of 40% of the time spent above the MIC of the bacteria in question (fT>MIC=40%) for a temocillin dose of 50mg/kg/day in 2 IV injections of 30 min spaced 12h apart, | 24 months
  Achievement of the theoretical PK/PD target of 40% of the time spent above the MIC of the bacteria in question (fT>MIC=40%) for a temocillin dose of 50mg/kg/day in 2 IV injections of 30 min spaced 12h apart, on the population modellisation of the unbound plasma concentration of temocillin over 24h. Samples taken 1 hour after the start of a temocillin infusion then between 6 and 8 hours after the start of the infusion or sample taken 2 hours after the start of a temocillin infusion then between 10 and 12 hours after the start of the infusion

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel LIGNIERES, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, Ap-hp / DRCI, France

IPD SHARING:
Plan to Share IPD: Undecided